CLINICAL TRIAL: NCT01460576
Title: Improving Prematurity-Related Respiratory Outcomes at Vanderbilt: The Prematurity and Respiratory Outcomes Program (PROP)
Brief Title: Improving Prematurity-Related Respiratory Outcomes at Vanderbilt
Acronym: IMPROV
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Paul Moore, Asscoc. Professor, Vanderbilt University Medical Center
Other Study IDs: 110833; 1U01HL101456 (NIH)
Record Dates: First submitted 2011-10-24; First posted 2011-10-27 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Preterm Birth; Bronchopulmonary Dysplasia; Chronic Lung Disease of Prematurity
Keywords: prematurity; respiratory disease; bronchopulmonary dysplasia
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva for DNA, plasma, red blood cells, urine and tracheal aspirates
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of IMPROV is to identify molecular mechanisms that contribute to lung injury and long-term breathing problems in preterm infants by investigating two interrelated biochemical pathways: the urea cycle-nitric oxide pathway and the glutathione pathway. The investigators hypothesize that prematurity-related limitations in the function of these important biochemical pathways contribute to respiratory disease risk over the first year of life.

DETAILED DESCRIPTION:
The primary goal of the IMPROV/PROP study is to identify biomarkers (biochemical, physiological and genetic) and clinical variables that are associated with and thus potentially predictive of pulmonary status in preterm infants at 1 year corrected age. IMPROV will test the hypothesis that biochemical immaturity and functional genetic variation in the urea cycle-nitric oxide (UC-NO) and glutathione (GSH) pathways influence the development and severity of bronchopulmonary dysplasia (BPD), a form of chronic lung disease that affects more than 10,000 premature infants each year in the US. IMPROV will also test the hypothesis that the duration and degree of NO insufficiency and free radical excess predicts BPD severity and correlates with persistence of lung problems after NICU discharge. Our hypothesis implicates (a) an immature liver and gastrointestinal ability to make citrulline and GSH, (b) inadequacy of nutritional amino acid substrate and (c) common genetic variations in the UC-NO and the GSH pathways in the pathogenesis of BPD. These factors limit the ability of the anatomically and functionally immature lung to respond to the physiologic and environmental stress of preterm birth. As part of the PROP multi-center study, novel approaches to characterizing lung status with non-invasive respiratory measures prior to NICU discharge will be employed. A composite primary outcome of morbidity that is based on serial parental reports of respiratory symptoms, medications, hospitalizations and dependence on technology during the first year of life has been developed.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are less than or equal to 7 days old;
* Gestational Age (GA) between 23 weeks and 0/7 days and 28 weeks and 6/7 days

Exclusion Criteria:

* The infant is not considered to be viable (decision made not to provide life-saving therapies);
* Congenital heart disease (not including PDA and hemodynamically insignificant VSD or ASD);
* Structural abnormalities of the upper airway, lungs or chest wall;
* Other congenital malformations or syndromes that adversely affect life expectancy or cardio-pulmonary development;
* Family is unlikely to be available for long-term follow-up.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted to the Neonatal Intensive Care Unit who are < 29 weeks gestational age
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2011-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Respiratory morbidity | one year corrected age
  Need for oxygen, respiratory medications, hospital admissions for respiratory disease or a positive response in at least 1 of 4 morbidity domains during at least 2 separate parental interviews.

SECONDARY OUTCOMES:
bronchopulmonary dysplasia | 36 weeks corrected age
  need for oxygen at 36 weeks based on a room air challenge

CONTACTS AND LOCATIONS:
Overall Officials: Judy L. Aschner, MD, Principal Investigator — Albert Einstein College of Medicine; Vanderbilt University School of Medicine
Locations (2):
- United States (2):
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vadivel A, Aschner JL, Rey-Parra GJ, Magarik J, Zeng H, Summar M, Eaton F, Thebaud B. L-citrulline attenuates arrested alveolar growth and pulmonary hypertension in oxygen-induced lung injury in newborn rats. Pediatr Res. 2010 Dec;68(6):519-25. doi: 10.1203/PDR.0b013e3181f90278. PMID 20805789
- [Background] Fike CD, Sidoryk-Wegrzynowicz M, Aschner M, Summar M, Prince LS, Cunningham G, Kaplowitz M, Zhang Y, Aschner JL. Prolonged hypoxia augments L-citrulline transport by system A in the newborn piglet pulmonary circulation. Cardiovasc Res. 2012 Aug 1;95(3):375-84. doi: 10.1093/cvr/cvs186. Epub 2012 Jun 6. PMID 22673370
- [Background] Ananthakrishnan M, Barr FE, Summar ML, Smith HA, Kaplowitz M, Cunningham G, Magarik J, Zhang Y, Fike CD. L-Citrulline ameliorates chronic hypoxia-induced pulmonary hypertension in newborn piglets. Am J Physiol Lung Cell Mol Physiol. 2009 Sep;297(3):L506-11. doi: 10.1152/ajplung.00017.2009. Epub 2009 Jul 17. PMID 19617312